CLINICAL TRIAL: NCT01837940
Title: Efficacy of a Dietary Supplementation With Lactobacillus Reuteri DSM 17938 for Digestive Health in an Elderly Population
Brief Title: Efficacy of a Dietary Supplementation With Lactobacillus Reuteri for Digestive Health in an Elderly Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Robert Brummer, Professor and Dean, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/309
Record Dates: First submitted 2013-03-26; First posted 2013-04-23 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Constipation; Diarrhea; Indigestion; Reflux; Abdominal Pain
MeSH Terms: conditions — Constipation; Diarrhea; Dyspepsia; Gastroesophageal Reflux; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- dietary supplement (Active Comparator): Lactobacillus reuteri DSM 17938
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938

INTERVENTIONS:
Dietary Supplement: Placebo — Galactooligosaccharide (GOS) and rhamnose in a powder formulation
  Arms: Placebo
Dietary Supplement: Lactobacillus reuteri DSM 17938 — Lactobacillus reuteri DSM17938, Galactooligosaccharide (GOS), rhamnose in a powder formulation
  Arms: dietary supplement

SUMMARY:
The purpose of this study is to investigate the effect of a daily supplement consisting of the probiotic bacteria, Lactobacillus reuteri, on the digestive health among persons 65 years and older.

DETAILED DESCRIPTION:
The overall purpose of the study is to investigate the effect of daily supplementation, during a three months period, of L. reuteri on digestive health in an elderly Swedish population, residing in the municipality of Örebro. In addition an extensive screening of the study population in regard of overall health status, functionality and well-being as well as the composition of the gut microbiome will be assessed prior study start through the collection of baseline data

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Informed consent signed by study participant or legal guardian

Exclusion Criteria:

* Known gastrointestinal disease, with strictures, malignance's and ischemia.
* Inflammatory bowel diseases (IBD)
* Participation in other clinical trials in the past three months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline Gastrointestinal symptoms to 3months | Baseline, at 2 months and at 3months/study end
  Gastrointestinal discomfort will be assessed through the gastrointestinal symptoms rating score (GSRS), a clinical rating scale for gastrointestinal symptoms. The GSRS includes 15 symptoms and uses a 7-point Likert scale in which 1 represents the most positive option and 7 the most negative.

SECONDARY OUTCOMES:
Change in use of intestinal motility regulating substances during the 3-month intervention period | at baseline and end of study ( 3months)
  Intestinal motility regulating substances (e.g anti-diarrheal and anti-constipation medication)

OTHER OUTCOMES:
Change in mood during the 3month intervention period | at baseline, 2months and 3monts/study end
  Mood changes will be assessed through the questionnaire hospital anxiety and depression scale (HADs)
Change in quality of life during the 3-month intervention period | at baseline, at baseline, 2months and 3monts/study end
  Quality of life will be assessed through the EuroQol questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan Brummer, MD, PhD, Principal Investigator — Örebro Universitet
Locations (1):
- Örebro University, Örebro, Närke, Sweden

REFERENCES:
- [Derived] Ostlund-Lagerstrom L, Kihlgren A, Repsilber D, Bjorksten B, Brummer RJ, Schoultz I. Probiotic administration among free-living older adults: a double blinded, randomized, placebo-controlled clinical trial. Nutr J. 2016 Sep 10;15(1):80. doi: 10.1186/s12937-016-0198-1. PMID 27612653